CLINICAL TRIAL: NCT00707083
Title: A Multicenter Study of Treatment Protocol for Childhood Acute Lymphoblastic Leukemia in China, 2008.
Brief Title: Two Combination Chemotherapy Regimens in Treating Children With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Kong Li, Dr., Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POWH-CRE-2008.077-T; CDR0000595184 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-06-27; First posted 2008-06-30 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; B-cell childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Dexamethasone; Mercaptopurine; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard- or Intermediate-Risk Maintenance Arm I (Active Comparator): Patients receive oral mercaptopurine and oral methotrexate on days 1-56, dexamethasone IV on days 1-5 and 29-33, vincristine IV on days 1 and 29, and methotrexate IT on day 50. Treatment repeats every 8 weeks for up to 8 (girls)-11 (boys) courses.
  Interventions: Drug: dexamethasone; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate
- Standard- or Intermediate-Risk Maintenance Arm II (Experimental): Patients receive oral mercaptopurine once daily on days 8-28 and 36-56; oral methotrexate once on days 8,15, 22, 36, 43, and 50; dexamethasone IV on days 1-5 and 29-33; and vincristine IV on days 1 and 29. Patients also receive methotrexate IT on day 1, every 8 weeks, for 8 courses.
  Interventions: Drug: dexamethasone; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate

INTERVENTIONS:
Drug: dexamethasone — Given oral
Drug: mercaptopurine — Given orally
Drug: methotrexate — Given orally
Drug: vincristine sulfate — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating acute lymphoblastic leukemia.

PURPOSE: This randomized clinical trial is studying the side effects of two combination chemotherapy regimens and to see how well they work in treating children with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of marrow suppression with 2 methods of maintenance treatment in children with acute lymphoblastic leukemia.
* Compare the incidence of liver toxicity with 2 methods of maintenance treatment in these patients.

Secondary

* Determine any difference in infection rates and related hospitalizations in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (high vs intermediate vs standard), age in years (0 to 5 vs 6 to 9 vs 10 to 17), and sex.

* Patients with standard-risk disease:

  * Induction therapy: Patients receive prednisolone IV or orally three times daily on days 1-7; oral dexamethasone three times daily on days 8-28; asparaginase IV over 1 hour or intramuscularly once on days 8, 11, 14, 17, 20, 23, 26, and 29; vincristine IV once on days 8, 15, 22, and 29; daunorubicin hydrochloride IV over 1 hour on days 8 and 15; and methotrexate intrathecally (IT) once on days 1, 15, and 33.
  * Early intensification (EI) therapy: Patients receive cyclophosphamide IV over 1 hour on day 36, cytarabine IV continuously on days 38-41 and 45-48, oral mercaptopurine once daily on days 36-50, and methotrexate IT on days 38 and 45.
  * Consolidation therapy: Two weeks after completing EI therapy, patients receive oral mercaptopurine once daily on days 1-56 and methotrexate IV over 24 hours and IT on days 8, 22, 36, and 50.
  * Delayed intensification (DI) therapy:

    * DI/a: Patients receive dexamethasone orally or IV three times daily on days 1-7 and 15-21, doxorubicin hydrochloride IV over 1 hour on days 1, 8, and 15; vincristine IV on days 1, 8, and 15; and asparaginase subcutaneously (SC) or IV over 1 hour on days 1, 4, 8, and 11.
    * DI/b: Patients receive cyclophosphamide IV over 1 hour on day 29, cytarabine IV continuously on days 31-34 and 38-41, oral thioguanine once daily on days 29-42, and methotrexate IT on days 31 and 38.
  * Maintenance therapy: Patients are randomized to one of two treatment arms. Patients who do not consent for randomization receive conventional therapy (arm I).

    * Arm I (conventional): Patients receive oral mercaptopurine and oral methotrexate on days 1-56, dexamethasone IV on days 1-5 and 29-33, vincristine IV on days 1 and 29, and methotrexate IT on day 50. Treatment repeats every 8 weeks for up to 8 courses for girls or 11 courses for boys.
    * Arm II (intervention): Patients receive oral mercaptopurine once daily on days 8-28 and 36-56; oral methotrexate once on days 8,15, 22, 36, 43, and 50; dexamethasone IV on days 1-5 and 29-33; and vincristine IV on days 1 and 29. Patients also receive methotrexate IT on day 1, every 8 weeks, for 8 courses.
* Patients with intermediate-risk disease:

  * Induction therapy: Patients receive prednisolone, dexamethasone, and asparaginase as in standard-risk induction therapy. Patients also receive vincristine IV and daunorubicin hydrochloride IV over 1 hour on days 8, 15, 22, and 29; methotrexate IT on day 1; and triple intrathecal therapy (TIT; high-dose methotrexate, cytarabine, hydrocortisone sodium succinate) on days 15 and 33.
  * First EI therapy: Patients receive cyclophosphamide, cytarabine, and mercaptopurine as in standard-risk EI. Patients also receive TIT on day 38.
  * Second EI therapy: Beginning 2 weeks after completing first EI, patients receive cyclophosphamide over 1 hour on day 1, oral mercaptopurine on days 1-14, cytarabine IV on days 3-6 and 10-13, and TIT on day 3.
  * Consolidation therapy: Beginning 2 weeks after completing second EI, patients receive mercaptopurine as in standard-risk consolidation therapy. Patients also receive methotrexate IV over 24 hours and TIT on days 8, 22, 36, and 50.
  * First DI therapy: Patients receive treatment as in standard-risk DI.
  * Interim maintenance therapy: Patients receive oral mercaptopurine and oral methotrexate on days 1-56.
  * Second DI therapy: Patients receive DI/a and D1/b (without methotrexate) as in standard-risk DI. Patients also receive TIT on days 31 and 38.
  * Maintenance therapy: Patients are randomized to 1 of 2 treatment arms:

    * Arm I (conventional): Patients receive mercaptopurine, methotrexate, dexamethasone, and vincristine as in standard-risk maintenance therapy arm I. Patients also receive TIT on day 50. Treatment repeats every 8 weeks for up to 8 courses for girls or 11 courses for boys.
    * Arm II (intervention): Patients receive treatment as in standard-risk maintenance therapy arm II.
* Patients with high-risk disease:

  * Induction therapy: Patients receive treatment as in intermediate-risk induction therapy.
  * First EI therapy: Patients receive treatment as in intermediate-risk first EI.
  * Second EI therapy: Patients receive treatment as in intermediate-risk second EI.
  * Consolidation therapy (interval between blocks is 2 weeks):

    * Block 1: Patients receive dexamethasone orally or IV three times daily on days 1-5, vincristine IV on days 1 and 6, high-dose methotrexate IV over 24 hours on day 1, cyclophosphamide IV over 1 hour twice daily on days 2-4, cytarabine IV over 3 hours twice on day 5, asparaginase IV over 2 hours on days 6 and 11, and TIT on day 1.
    * Block 2: Patients receive dexamethasone, high-dose methotrexate, asparaginase, and TIT as in block 1. Patients also receive vindesine IV twice daily on days 1 and 6, ifosfamide IV over 1 hour twice daily on days 2-4, and daunorubicin hydrochloride IV over 24 hours on day 5.
    * Block 3: Patients receive dexamethasone and asparaginase as in block 1. Patients also receive high-dose cytarabine IV over 3 hours twice daily on days 1 and 2, etoposide IV over 1 hour five times on days 3-5, and TIT on day 5.
  * Blocks 1-3 are then repeated once. Patients then proceed to delayed intensification therapy.
  * Delayed intensification therapy: Patients receive dexamethasone orally or IV three times daily on days 1-7 and 15-21; doxorubicin hydrochloride IV and vincristine IV on days 8, 15, 22, and 29; and asparaginase IV on days 8, 11, 15, and 18. Patients also receive cyclophosphamide IV on day 36, cytarabine IV on days 38-41 and 45-48, thioguanine IV on days 36-49, and TIT on days 38 and 45.
  * Maintenance therapy: Patients receive oral mercaptopurine and oral methotrexate once daily on days 1-14, cyclophosphamide over 1 hour and cytarabine over 1 hour once between days 15-21, oral dexamethasone two or three times daily for 5 days between days 29-35, vincristine IV on day 29, and TIT on day 22. Treatment repeats every 4 weeks. After 10 courses, patients no longer receive TIT. After 12 courses, patients no longer receive cyclophosphamide and cytarabine. At this time patients continue mercaptopurine and methotrexate on days 1-21. After 20 courses, patients no longer receive dexamethasone or vincristine. At this time, patients continue mercaptopurine and methotrexate on days 1-28. Females receive up to 17 courses and males up to 23 courses.

Some patients may also undergo radiotherapy or stem cell transplantation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia meeting 1 of the following risk definitions:

  * Standard-risk disease:

    * Age 1 to 9 years
    * White blood cell (WBC) < 50/mm^3 OR t(12;21) or molecular fusion product -positive disease
    * Good response to prior prednisone (day 8 peripheral blood blast < 1,000/mm^3)
    * None of the following subtypes:

      * T-cell
      * t(9;22)
      * t(4;11)
      * t(1;19)
      * Molecular
    * Bone marrow (BM) M1 or M2 on day 15, BM remission (< 5% blast) on day 33
  * Intermediate-risk disease:

    * Good response to prior prednisone
    * BM M1/M2 on day 15
    * Meets 1 of the following criteria:

      * At least 10 years old
      * WBC > 50/mm^3
      * Under 1 year old without Mixed Lineage Leukemia (MLL) gene rearrangement
      * T-cell OR t(1;19) or molecular fusion product positive.
      * Standard-risk patient with BM M3 on day 15
      * If minimal residual disease (MRD) available, day 33 MRD < 10^-2
  * High-risk disease, meeting 1 of the following criteria:

    * Poor response to prior prednisone
    * t(9;22) or molecular fusion product (BCR/ABL1), t(4;11) or molecular fusion product (MLL/AF4)
    * Intermediate-risk patient with BM M3 on day 15
    * BM M2/M3 on day 33
    * If MRD available, flow cytometry/polymerase chain reaction (PCR) > 10% on days 15 OR MRD > 10^-2 on day 33 OR MRD (before mini-M phase or M phase) > 10^-3 on day 84

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2231 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Bone marrow suppression and liver toxicity | 24 or 30 months of chemotherapy
  compare marrow suppression in the two arms of maintenance treatment

SECONDARY OUTCOMES:
overall and event-free survival | 3 years after stop treatment
Hospitalization rate during maintenance treatment | 24 or 30 months after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Kong Li, MD, Principal Investigator — Prince of Wales Hospital
Locations (2):
- China (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital - Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, Zou Y, Chen X, Wang S, Guo Y, Yang W, Zhang L, Chen Y, Zhang Y, Zhu X. Minimal residual disease surveillance at day 90 predicts long-term survival in pediatric patients with T-cell acute lymphoblastic leukemia. Leuk Lymphoma. 2020 Dec;61(14):3460-3467. doi: 10.1080/10428194.2020.1805739. Epub 2020 Aug 11. PMID 32779947
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00707083